CLINICAL TRIAL: NCT06914466
Title: Neural Mechanisms and Clinical Applications of Deep Brain Stimulation for Modulating Sleep Dysregulation in Parkinson's Disease
Brief Title: Neural Mechanisms and Clinical Applications of DBS for Modulating Sleep Dysregulation in PD
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 20250322
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Deep Brain Stimulation; Parkinson's Disease and Parkinsonism; Sleep Disorder
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Sleep Wake Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep Brain Stimulation

SUMMARY:
Parkinson's disease (PD) is a prevalent neurodegenerative disorder characterized by both motor and non-motor symptoms. Subthalamic nucleus (STN) deep brain stimulation (DBS) effectively alleviates motor symptoms; however, non-motor symptoms such as sleep disorders significantly impair patients' quality of life. While preliminary evidence suggests DBS may improve sleep, the underlying neural mechanisms and long-term effects on sleep regulation remain poorly elucidated. This study employs a wearable polysomnography (PSG) device to investigate how STN-DBS modulates sleep architecture, local field potentials (LFPs), and clinical outcomes in PD patients. We hypothesize that STN-DBS contributes to both the regulation and disruption of normal sleep behavior. By synchronizing PSG with STN-LFP recordings under DBS-ON and DBS-OFF conditions, we aim to decode sleep stages using STN-LFPs, characterize PD-specific sleep abnormalities (e.g., sleep architecture, atonia), and analyze DBS-induced LFP changes and their correlations with clinical efficacy. According to the above data, the sleep stage characteristics were decoded, and the algorithm was used to determine the optimal clinical threshold current amplitude to improve sleep. Then, the patients will be given adaptive stimulation, and the sleep quality was monitored to verify its efficacy.This study will provide a neurophysiological foundation for developing closed-loop stimulation strategies targeting sleep dysfunction in PD.

DETAILED DESCRIPTION:
This single-center longitudinal observational study will enroll 20 idiopathic Parkinson's disease (PD) patients with bilateral subthalamic nucleus (STN) deep brain stimulation (DBS) systems (Medtronic Percept™ PC) to evaluate the neurophysiological mechanisms of DBS in sleep regulation. Participants will undergo preoperative clinical assessments (MDS-UPDRS III for motor symptoms, NMSS for non-motor symptoms, PDSS for sleep-specific dysfunction) and two nights of wearable PSG recordings. Postoperatively, DBS parameters will be optimized at 1 month for motor symptom control. Follow-up evaluations at 3, 6, and 12 months post-operation include in-hospital PSG and local field potential (LFP) recordings: Night 1 captures data under DBS-OFF conditions, followed by Night 2 with DBS-ON under optimized programming, alongside repeated clinical assessments. Sleep architecture (NREM/REM stages, arousal indices,atonia) and STN-LFPs will be analyzed and correlated with clinical outcomes. Machine learning models will identify LFP biomarkers predictive of sleep improvement to inform closed-loop stimulation strategies. Based on the machine learning results, we will investigate the adaptive algorithm and validate its effectiveness in the second phase. Adaptive stimulation will be administered for one month, followed by two consecutive nights of polysomnography (PSG) monitoring and Parkinson's Disease Sleep Scale (PDSS) assessments at the study interval endpoint. Subsequently, patients will undergo routine open-loop stimulation for one month, with two additional consecutive nights of PSG monitoring and PDSS evaluations conducted upon completion of this phase. Sleep improvement outcomes will be systematically compared between the two stimulation modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease: The diagnostic criteria for Parkinson's disease are the Clinical Diagnostic Criteria of UK PD Society Brain Bank Clinical Diagnostic Criteria or 2015 MDS Clinical Diagnostic Criteria for PD.All diagnoses of Parkinson's disease were made by three neurologists who were experienced in the field of movement disorders.
2. Patients who underwent bilateral STN-DBS(Medtronic Percept™ PC)
3. Patients who can cooperate with the completion of postoperative follow-up and clinical evaluation.

Exclusion Criteria:

1. Patients who underwent other brain surgery;
2. Other patients with secondary Parkinson's syndrome and Parkinsonism-plus syndrome;
3. Patients with other central nervous system and peripheral nervous system diseases;
4. Patients complicated with severe medical system diseases, or unable to tolerate clinical evaluation;
5. Patients with severe mental illness;
6. Patients who cannot complete informed consent due to cognitive and communication barriers, or refuse to sign informed consent.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who 2.underwent bilateral STN-DBS(Medtronic Percept™ PC) and consent to participate in the sleep study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of REM sleep stage | 12 months
  Sleep fragmentation frequency and duration will be measured using PSG
Subjective Sleep Quality | 12 months
  Change in subjective sleep quality will be measured between the different conditions. The measure will be captured using the Parkinson's disease sleep scale, PDSS.

CONTACTS AND LOCATIONS:
Overall Officials: yuqing Zhang, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China